CLINICAL TRIAL: NCT05525234
Title: A Prospective, Randomized, Double-blind, Placebo-controlled Study of Thalidomide in the Treatment of Refractory Uremic Pruritus
Brief Title: A Study of Thalidomide in the Treatment of Refractory Uremic Pruritus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022.06.15
Record Dates: First submitted 2022-08-29; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Haemodialysis; Uremic Pruritus; Thalidomide
MeSH Terms: interventions — Thalidomide

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thalidomide group (Experimental): Thalidomide tablets, 50mg/day, increase or decrease dose according to itch score. The maximum dose is 100mg/day.
  Interventions: Drug: Thalidomide
- Placebo group (Placebo Comparator): Palacebo tablets, 50mg/day, increase or decrease dose according to itch score. The maximum dose is 100mg/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thalidomide — Start with oral thalidomide at 50mg/day, increase or decrease the dose according to itching relief, the maximum dose is 100mg/day
  Arms: Thalidomide group
Drug: Placebo — Start with oral placebo at 50mg/day, increase or decrease the dose according to itching relief, the maximum dose is 100mg/day
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of thalidomide in the treatment of refractory uremic pruritus in maintenance hemodialysis patients.

DETAILED DESCRIPTION:
A prospective, randomized, double-blind, placebo-controlled study was conducted to explore the efficacy and safety of thalidomide in the treatment of refractory urmia pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis patients (≥3 month), 3 times/week, 4 hours/session
* spKT/V≥1.2
* The diagnosis was refractory urmia pruritus and pruritus score ≥8 score
* Patients with sleep disorders need to stop sleeping pills
* Be able to complete the form by yourself or with the help of others
* Informed consent

Exclusion Criteria:

* Participants in other clinical trials within 1 month
* People with thalidomide allergy
* Accompanied by severe calcium and phosphorus metabolism disorder (serum calcium≥3.0mmol/L or Serum phosphorus≥2.8mmol/L or Serum iPTH≥800pg/mL)
* Patients with other medical conditions that cause itchy skin
* With severe systemic infection, severe anemia and other serious complications
* Patients with peripheral neuropathy
* Other serious systemic diseases include systemic lupus erythematosus, multiple myeloma, thrombotic microangiopathy, and extensive metastasis of malignant tumors
* Patients with a history of thromboembolism were excluded from PICC-induced thrombosis
* Pregnant woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Pruritus score | 12 weeks
  Comparison of pruritus score between treatment group and control group at 12 weeks

SECONDARY OUTCOMES:
Efficacy index and response rate | 12 weeks
  Comparison of efficacy index and response rate between treatment group and control group. Efficacy index (%)=(Total score before treatment-Total score after treatment）/Total score before treatment×100%, Response rate: Efficacy index ≥30% is effective; Efficacy index <30% is noneffective.
Pittsburgh sleep quality score | 12 weeks
  Comparison of Pittsburgh sleep quality score between treatment group and control group

OTHER OUTCOMES:
Security Index | 12 weeks
  Comparison of vital signs including breathing (breaths per minute), heart rate (beats per minute), blood pressure (mmHg), laboratory tests including white blood cell count (×109/L), hemoglobin (g/L), alanine transaminase (IU/L), aspertate Aminotransferase(IU/L), blood glucose (mmol/L), albumin (g/L), high sensitivity C-reactive protein (mg/L) and so on and severity of adverse events assessed according to CTC-AE 4.0 criteria between the treatment and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Renhua Lu, Doctor, Principal Investigator — Ren Ji Hospital, School of Medicine Shanghai Jiao Tong University